CLINICAL TRIAL: NCT00392925
Title: A Phase 2A, Randomized, Controlled, Double-Blind, Multicenter Study to Evaluate the Safety, Tolerability, and Effect on Body Weight of Recombinant-Methionyl Human Leptin Administered in Conjunction With Pramlintide in Overweight and Obese Subjects
Brief Title: A Study to Evaluate the Effect on Body Weight of Leptin Administered in Conjunction With Pramlintide in Overweight and Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFA101
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; pramlintide; leptin; Amylin
MeSH Terms: conditions — Overweight; Obesity | interventions — pramlintide; metreleptin; recombinant methionyl human leptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo and Metreleptin (Experimental): Placebo-pramlintide 600 microliters (µL) twice a day (BID) and metreleptin (recombinant-methionyl human leptin) 5 milligram (mg) BID, 20 weeks
  Interventions: Drug: metreleptin; Drug: placebo-pramlintide 600 uL
- Pramlintide Acetate and Placebo (Experimental): Lead-in period: 2 weeks pramlintide acetate 180 mcg BID, then 2 weeks pramlintide acetate 360 mcg BID Study period: Pramlintide acetate 360 mcg BID and placebo-metreleptin 1 mL BID, 20 weeks
  Interventions: Drug: pramlintide acetate 360 mcg; Drug: placebo-metreleptin 1 mL
- Pramlintide Acetate and Metreleptin (Experimental): Lead-in period: 2 weeks pramlintide acetate 180 mcg BID, then 2 weeks pramlintide acetate 360 mcg BID Study period: Pramlintide acetate 360 mcg BID and metreleptin (recombinant-methionyl human leptin) 5 mg BID, 20 weeks
  Interventions: Drug: pramlintide acetate 360 mcg; Drug: metreleptin
- Lead-In Period (Other): During the Lead-In Period before a participant was randomized to a study arm, the participant received 180 mcg pramlintide acetate twice a day (BID) for 2 weeks, followed by 360 mcg pramlintide acetate BID for 2 weeks (total of 4 weeks in the Lead-In Period).
  Interventions: Drug: pramlintide acetate 360 mcg; Drug: Pramlintide acetate 180 mcg

INTERVENTIONS:
Drug: pramlintide acetate 360 mcg — subcutaneous injection, twice a day, 360mcg
  Other Names: SYMLIN®
  Arms: Lead-In Period; Pramlintide Acetate and Metreleptin; Pramlintide Acetate and Placebo
Drug: metreleptin — subcutaneous injection, twice a day, 5mg
  Other Names: recombinant-methionyl human leptin
  Arms: Placebo and Metreleptin; Pramlintide Acetate and Metreleptin
Drug: placebo-pramlintide 600 uL — twice a day
  Arms: Placebo and Metreleptin
Drug: placebo-metreleptin 1 mL — twice a day
  Arms: Pramlintide Acetate and Placebo
Drug: Pramlintide acetate 180 mcg — subcutaneous injection twice a day, 180 mcg
  Other Names: SYMLIN®
  Arms: Lead-In Period

SUMMARY:
This study will evaluate the safety, tolerability, and effect on body weight of leptin, injected subcutaneously, in combination with pramlintide, injected subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* Is obese (Body Mass Index [BMI]>=30kg/m^2 and <=35kg/m^2); or overweight (BMI>=27kg/m^2 and <30kg/m^2) with abdominal obesity, based on the following: *waist circumference >102 cm if male, *waist circumference >88 cm if female
* Is a nonsmoker (has not smoked for at least 6 months prior to the study)
* Consumes a morning and evening meal each day

Exclusion Criteria:

* Is diagnosed with type 2 diabetes
* Is currently enrolled or plans to enroll in a diet, weight loss, or exercise program with the specific intent of losing weight (subjects who have been following an exercise regimen resulting in stable weight maintenance for at least 2 months prior to enrollment are eligible for study inclusion)
* Has been treated over the past 2 months, is currently treated, or is expected to require or undergo treatment with any of the following medications: *antiobesity agents (prescription or over-the-counter), *antipsychotic agents, *antiepileptic agents, *antidepressant agents, *drugs that directly affect gastrointestinal motility
* Has received any investigational drug within 30 days or within a period corresponding to 5 half-lives of that drug, whichever is greater, prior to this study starting
* Has previously received treatment with recombinant leptin or pramlintide

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (12):
- United States (12):
  - Research Site, DeLand, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Butte, Montana
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Salt Lake City, Utah
  - Research Site, Olympia, Washington

REFERENCES:
- [Derived] Chan JL, Koda J, Heilig JS, Cochran EK, Gorden P, Oral EA, Brown RJ. Immunogenicity associated with metreleptin treatment in patients with obesity or lipodystrophy. Clin Endocrinol (Oxf). 2016 Jul;85(1):137-49. doi: 10.1111/cen.12980. Epub 2016 Feb 2. PMID 26589105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 October 2006 started Lead-in Period. 20 September 2007 final visit. Study conducted at clinics with obese patients (body mass index [BMI]greater than, equal to [≥]30 to less than, equal to [≤]35 kg/m^2) or overweight patients (BMI ≥27 to <30 kg/m^2) and abdominal obesity = waist circumference >102 centimeters (cm) for males; >88 cm for females.
Pre-assignment Details: 177 participants enrolled into single blind lead-in period with pramlintide treatment and a diet, 38 withdrew before double blind randomization into 1 of 3 treatment arms. Participants who lost between 2% and 8% of their enrollment body weight during the lead-in period were randomized at Visit 4 (baseline/Day 1) to 1 of 3 treatment groups.
Groups:
- Non-Randomized From 4 Week Lead-In: During the 4-week lead-in period, all participants self administered a subcutaneous injection of pramlintide acetate 180 mcg twice per week (BID) for 2 weeks followed by pramlintide 360 mcg BID for 2 weeks while following a diet aimed at creating a 40% caloric deficit relative to their estimated weight-maintenance energy needs. Participants who lost between 2% and 8% of their enrollment body weight during the lead-in period were randomized at Visit 4 (baseline/Day 1) to 1 of 3 treatment groups (metreleptin, pramlintide, or pramlintide+metreleptin). 38 participants were not Randomized into one of the 3 treatment groups and withdrew from the study.
- Metreleptin: Participants self administered subcutaneous (SC) injections of Placebo matched to pramlintide (Placebo-P) BID plus Metreleptin 5 milligram (mg) BID. Dosing for up to 20 weeks. Participants were asked to maintain a 20% caloric deficit during the treatment period.
- Pramlintide Acetate: Participants self administered subcutaneous (SC) injections of Pramlintide acetate 360 mcg BID plus Placebo matched to Metreleptin (Placebo-M) BID. Dosing for up to 20 weeks. Participants were asked to maintain a 20% caloric deficit during the treatment period.
- Pramlintide Acetate + Metreleptin: Participants self administered subcutaneous (SC) injections of Pramlintide acetate 360 mcg BID plus Metreleptin 5 mg BID. Dosing for up to 20 weeks. Participants were asked to maintain a 20% caloric deficit during the treatment period.
Period: 4 Week Lead-In Period - Non-Randomized
Arm/Group | Non-Randomized From 4 Week Lead-In | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Started | 177 | 0 | 0 | 0
Completed | 139 | 0 | 0 | 0
Not Completed | 38 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0 | 0
Not completed — did not meet weight loss criteria | 16 | 0 | 0 | 0
Period: Randomization to Treatment Group Period
Arm/Group | Non-Randomized From 4 Week Lead-In | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Started | 0 | 27 | 56 | 56
Completed | 0 | 19 (AT Week 20) | 37 (At Week 20) | 38 (At Week 20)
Not Completed | 0 | 8 | 19 | 18
Not completed — Withdrawal by Subject | 0 | 2 | 6 | 8
Not completed — Adverse Event | 0 | 3 | 3 | 5
Not completed — Protocol Violation | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 3 | 8 | 4

BASELINE CHARACTERISTICS:
Population: 177 participants enrolled into the study and started a 4 week lead-in period. 38 participants withdrew from the study during the lead-in period and 139 participants were randomized into one of 3 treatment groups. Baseline demographics presented for all 177 enrolled participants, by treatment group or those not randomized to a treatment group.
Groups:
- Metreleptin: Participants self administered subcutaneous (SC) injections of Placebo matched to pramlintide (Placebo-P) BID plus Metreleptin 5 mg BID. Dosing for up to 20 weeks. Participants were asked to maintain a 20% caloric deficit during the treatment period.
- Non-Randomized From 4 Week Lead-In: During the 4-week lead-in period, all participants self administered subcutaneous (SC) injections of pramlintide acetate 180 mcg twice per week (BID) for 2 weeks followed by pramlintide acetate 360 mcg BID for 2 weeks while following a diet aimed at creating a 40% caloric deficit relative to their estimated weight-maintenance energy needs. Participants who lost between 2% and 8% of their enrollment body weight during the lead-in period were randomized at Visit 4 (baseline/Day 1) to 1 of 3 treatment groups (metreleptin, pramlintide, or pramlintide+metreleptin). 38 participants were not randomized into one of the 3 treatment groups and withdrew from the study.
- Total: Total of all reporting groups
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin | Non-Randomized From 4 Week Lead-In | Total
Number analyzed (Participants) | 27 | 56 | 56 | 38 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (8.06) | 38.3 (9.13) | 38.5 (8.42) | 37.9 (7.51) | 38.6 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 35 | 35 | 24 | 111
  Male | 10 | 21 | 21 | 14 | 66
Region of Enrollment [Number; unit: participants]
  United States | 27 | 56 | 56 | 38 | 177
Body Weight at Enrollment [Mean (Standard Deviation); unit: kg] — Body weight was measured in kilograms (kg) at enrollment, Visit 2 (Week -4).
  kg | 93.80 (14.322) | 91.70 (11.085) | 93.89 (12.834) | 94.54 (16.027) | 93.32 (13.246)
Body Weight at Baseline [Mean (Standard Deviation); unit: kg] — Body weight was measured in kg at Day 1, baseline for randomized participants.
  kg | 89.83 (13.389) | 88.05 (10.507) | 89.88 (12.355) | NA (NA) — Non-randomized participants are not included in the Baseline Weight because they did not reach Day 1 baseline. They withdrew from the study before randomization. | 89.13 (11.807)
Body Mass Index (BMI) at Enrollment [Mean (Standard Deviation); unit: kg/m^2] — BMI was measured as kilogram per meter of height squared (kg/m^2).
  kg/m^2 | 32.0 (2.15) | 31.5 (2.03) | 32.0 (2.10) | 32.5 (1.95) | 32.0 (2.07)

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Change From Baseline to Week 16 in Body Weight - Evaluable Population
Description: Absolute change in body weight as measured in kilograms (kg) from baseline to Week 16. Baseline defined as Day 1 of randomized treatment.
Time Frame: Baseline to Week 16
Population: Evaluable: randomized participants with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with the protocol as per the sponsor. Participants excluded from the Evaluable Population were identified prior to the unblinding process. n=number with non-missing body weight data at Week 16 in each treatment group.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
kg | -2.68 (0.952) | -3.30 (0.698) | -6.46 (0.682)
Statistical Analysis 1: Comparison: Pramlintide Acetate vs Pramlintide Acetate + Metreleptin; Based on an Analysis of Covariance model including factors for treatment group, sex, enrollment body mass index (BMI) category, lead-in body weight loss category, and baseline (Day 1) weight as a covariate. The p-value is for testing the null hypothesis of no difference between treatments. Analysis performed two-sided at a 5% significance level to compare treatment groups; Test type: Superiority or Other; p = 0.0004, ANCOVA

2. Secondary Outcome: LS Mean Percent Change in Body Weight From Baseline to Weeks 4, 8, 12, 16, and 20 - Evaluable Population
Description: Least Squares (LS) mean percent change in body weight from baseline to Weeks 4 through 20. Baseline defined as Day 1 of randomized treatment.
Time Frame: Baseline up to Week 20
Population: Evaluable: randomized with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with protocol (per sponsor). Those excluded were identified prior to the unblinding process. n=number with non-missing body weight data (at visit) in each treatment group.
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
percentage of change
  Week 4 (n=19, 38, 36) | -0.70 (0.429) | -1.55 (0.310) | -2.36 (0.311)
  Week 8 (n=19, 38, 36) | -2.08 (0.591) | -2.74 (0.427) | -4.81 (0.429)
  Week 12 (n=19, 38, 36) | -3.17 (0.796) | -3.39 (0.575) | -6.13 (0.577)
  Week 16 (n=19, 38, 36) | -3.37 (1.025) | -3.85 (0.740) | -7.59 (0.743)
  Week 20 (n=19, 37, 36) | -3.62 (1.277) | -3.89 (0.925) | -8.21 (0.926)

3. Secondary Outcome: LS Mean Absolute Change From Baseline to Weeks 4, 8, 12, 20 in Body Weight - Evaluable Population
Description: Least Squares (LS) mean absolute change in body weight as measured in kilograms (kg) from baseline to Weeks 4, 8, 12, 20. Baseline defined as Day 1 of randomized treatment
Time Frame: Baseline to Week 20
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
kg
  Week 4 (n=19, 38, 36) | -0.66 (0.387) | -1.43 (0.284) | -2.13 (0.277)
  Week 8 (n=19, 38, 36) | -1.66 (0.540) | -2.32 (0.396) | -4.16 (0.387)
  Week 12 (n=19, 38, 36) | -2.59 (0.742) | -2.97 (0.544) | -5.28 (0.532)
  Week 20 (n=19, 37, 36) | -2.80 (1.199) | -3.30 (0.881) | -6.90 (0.859)

4. Secondary Outcome: LS Mean Absolute Change in Body Weight From Enrollment to Weeks 4, 8, 12, 16, and 20 - Evaluable Population
Description: Least Squares (LS) mean change in body weight as measured in kilograms (kg) from enrollment to each study visit. Enrollment was Visit 2 (Week -4) which was the start of the Lead-In Period. After the 4 week Lead-In Period, at Day 1, the participant was randomized to one of the 3 study arms and the participant was treated as per that arm up to Week 20.
Time Frame: Enrollment to Week 20
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kg
Groups:
- Pramlintide + Metreleptin: Participants self administered subcutaneous (SC) injections of Pramlintide 360 mcg BID plus Metreleptin 5 mg BID. Dosing for up to 20 weeks. Participants were asked to maintain a 20% caloric deficit during the treatment period.
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
kg
  Week 4 (n=19, 38, 36) | -5.22 (0.483) | -5.93 (0.353) | -6.72 (0.346)
  Week 8 (n=19, 38, 36) | -6.25 (0.635) | -6.85 (0.464) | -8.77 (0.455)
  Week 12 (n=19, 38, 36) | -7.18 (0.822) | -7.50 (0.60) | -9.89 (0.590)
  Week 16 (n=19, 38, 36) | -7.28 (1.028) | -7.84 (0.751) | -11.07 (0.737)
  Week 20(n=19, 37, 36) | -7.41 (1.262) | -7.86 (0.923) | -11.52 (0.904)

5. Secondary Outcome: LS Mean Percent Change in Body Weight From Enrollment to Weeks 4, 8, 12, 16, and 20 - Evaluable Population
Description: Least Squares (LS) mean percent change is percentage that body weight changed over time at each visit. Enrollment was Visit 2 (Week -4) which was the start of the Lead-In Period. After the 4 week Lead-In Period, at Day 1, the participant was randomized to one of the 3 study arms and treated up to Week 20.
Time Frame: Enrollment to Week 20
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
percentage of change
  Week 4 (n=19, 38, 36) | -5.46 (0.512) | -6.20 (0.369) | -7.18 (0.371)
  Week 8 (n=19, 38, 36) | -6.77 (0.654) | -7.33 (0.473) | -9.50 (0.474)
  Week 12 (n=19, 38, 36) | -7.80 (0.836) | -7.95 (0.604) | -10.75 (0.606)
  Week 16 (n=19, 38, 36) | -7.99 (1.058) | -8.37 (0.764) | -12.13 (0.767)
  Week 20 (n=19, 37, 36) | -8.22 (1.286) | -8.42 (0.931) | -12.72 (0.932)

6. Secondary Outcome: Initial, Late, and Overall Rates of LS Mean Absolute Change in Body Weight From Day 1 to Week 20 - Evaluable Population
Description: Initial (Day 1 through Week 12), late (Week 12 through Week 20), and overall (Day 1 through Week 20) rates of Least squares (LS) mean absolute change in body weight were defined by the slopes of the regression lines fitted to the observed body weights during the periods from Baseline (Day 1) through each visit to Week 20. Initial, late and overall absolute change was measured in kilograms of body weight per week (kg/week). Baseline refers to Visit 4 (Day 1 of randomization period).
Time Frame: Baseline to Week 20
Population: Evaluable: randomized with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with protocol (per sponsor). Those excluded were identified prior to the unblinding process.
Measure: Least Squares Mean (Standard Error); unit: kg/week
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
kg/week
  Initial rate of absolute change | -0.23 (0.060) | -0.25 (0.044) | -0.46 (0.043)
  Late rate of absolute change | -0.02 (0.079) | -0.05 (0.058) | -0.20 (0.057)
  Overall rate of absolute change | -0.16 (0.059) | -0.17 (0.043) | -0.36 (0.042)

7. Secondary Outcome: Number of Participants Achieving at Least 5% and at Least 10% Body Weight Loss From Baseline to Weeks 16 and 20, and Number of Participants With Sustained Weight Loss in Each Category - Evaluable Population
Description: Baseline refers to Visit 4 (Day 1 of randomization period). Number of participants with 5% or more and 10% or more change in weight from baseline at each visit. Number of participants with 5% or more change in weight that was sustained through Week 16. Number of participants with 10% or more change in weight that was sustained through Week 20.
Time Frame: Baseline to Weeks 16 and Weeks 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
participants
  Weight Loss of 5% or more Week 16 (n=19, 38, 36) | 5 | 13 | 22
  Weight Loss of 5% or more Week 20(n=19, 37, 36) | 6 | 14 | 25
  5% Loss Week 16 Sustained (n=19, 38, 36) | 5 | 12 | 21
  Weight Loss of 10% or more Week 16(n=19, 38, 36) | 1 | 1 | 9
  Weight Loss of 10% or more Week 20(n=19, 37, 36) | 2 | 2 | 11
  10% Loss Week 16 Sustained (n=19, 38, 36) | 1 | 1 | 9

8. Secondary Outcome: LS Mean Percent Change in Weight From Enrollment to Baseline and LS Mean Percent Change in Excess Weight From Enrollment to Baseline - Evaluable Population
Description: Excess body weight: the difference between a participant's actual body weight and the weight a participant of his/her height would have if his/her BMI were 24.9 kg/m2. Excess body weight at a given visit was calculated as body weight in kilograms (kg) at that visit minus 24.9 × height in meters (m)^2 or 0, whichever was greater. If a participant achieved a normal BMI (24.9 kg/m^2), that subject was considered to have no excess weight. Additional weight loss that occurred after a normal BMI was achieved was not included in the calculation of excess weight loss. Enrollment was Visit 2 (Week -4), the start of the Lead-In Period. Baseline was Day 1 of the randomization to a study arm.
Time Frame: Enrollment to Baseline
Population: Evaluable: randomized with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with protocol (per sponsor). Those excluded were identified prior to the unblinding process. Number with non-missing body weight data at Day 1 of Randomization were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Groups:
- Lead-In Participants Randomized to Treatment on Day 1: During the 4-week lead-in period, all participants self administered subcutaneous (SC) injections of pramlintide 180 mcg twice per week (BID) for 2 weeks followed by pramlintide 360 mcg BID for 2 weeks while following a diet aimed at creating a 40% caloric deficit relative to their estimated weight-maintenance energy needs. Participants who lost between 2% and 8% of their enrollment body weight during the lead-in period were randomized at Visit 4 (baseline/Day 1) to a treatment group.
Arm/Group | Lead-In Participants Randomized to Treatment on Day 1
Number analyzed (Participants) | 93
percentage of change
  Percent Change in Weight from Enrollment | -4.42 (0.171)
  Percent Change in Excess Weight from Enrollment | -25.24 (1.085)

9. Secondary Outcome: LS Mean Absolute Change in Waist Circumference From Enrollment to Weeks 4, 8, 12, 16, 20 - Evaluable Population
Description: Waist circumference was measured in centimeters (cm). Least Squares mean = LS mean. Enrollment was Visit 2 (Week -4) which was the start of the 4 week Lead-In Period. At Day 1, the participant was randomized to one of the 3 study arms and the participant was treated up to Week 20.
Time Frame: Enrollment to Week 20
Population: Evaluable: randomized participants with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with the protocol (per sponsor). Those excluded from Evaluable were identified prior to unblinding. n=number with non-missing anthropometric data at visit in each treatment group.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
cm
  Week 4 (n=19, 38, 36) | -5.49 (0.940) | -6.78 (0.679) | -7.28 (0.682)
  Week 8 (n=19, 38, 36) | -5.74 (0.974) | -7.76 (0.703) | -8.75 (0.706)
  Week 12 (n=19, 38, 36) | -7.06 (1.077) | -8.46 (0.778) | -9.88 (0.782)
  Week 16 (n=19, 38, 36) | -6.84 (1.281) | -9.00 (0.925) | -10.66 (0.929)
  Week 20 (n=19, 37, 36) | -7.99 (1.509) | -9.17 (1.092) | -11.61 (1.094)

10. Secondary Outcome: LS Mean Absolute Change in Waist Circumference From Baseline to Weeks 4, 8, 12, 16, 20 - Evaluable Population
Description: Baseline was Visit 4 (Day 1 of randomization period). Waist circumference was measured in centimeters (cm).
Time Frame: Baseline to Week 20
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
cm
  Week 4 (n=19, 38, 36) | -1.08 (0.868) | -2.55 (0.626) | -2.95 (0.630)
  Week 8 (n=19, 38, 36) | -1.29 (0.833) | -3.51 (0.601) | -4.39 (0.605)
  Week 12 (n=19, 38, 36) | -2.63 (0.941) | -4.22 (0.679) | -5.54 (0.683)
  Week 16 (n=19, 38, 36) | -2.40 (1.177) | -4.75 (0.849) | -6.30 (0.854)
  Week 20 (n=19, 37, 36) | -3.60 (1.421) | -4.90 (1.029) | -7.28 (1.031)

11. Secondary Outcome: LS Mean Absolute Change in Hip Circumference From Screening up to Week 20 - Evaluable Population
Description: Screening (Week -5 or -6) was the first visit for a participant. This first visit determined participant eligibility and occurred prior to enrollment (Week -4). Hip circumference was measured in centimeters (cm).
Time Frame: Screening up to Week 20
Population: Evaluable: randomized participants with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with the protocol as per the sponsor. Those excluded from the Evaluable Population were identified prior to the unblinding process. Number with non-missing anthropometric data in each treatment group were analyzed.
Measure: Least Squares Mean (Standard Error); unit: cm
Groups:
- Pramlintide Acetate+ Metreleptin: Participants self administered subcutaneous (SC) injections of Pramlintide acetate 360 mcg BID plus Metreleptin 5 mg BID. Dosing for up to 20 weeks. Participants were asked to maintain a 20% caloric deficit during the treatment period.
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate+ Metreleptin
Number analyzed (Participants) | 19 | 37 | 36
cm | -6.36 (1.475) | -8.07 (1.082) | -10.27 (1.070)

12. Secondary Outcome: Number of Participants With BMI Change From Enrollment to Week 16 - Evaluable Population
Description: BMI was measured as kilogram per meter of height squared (kg/m^2). Enrollment was Visit 2 (Week -4). Participants who were obese (BMI of 30 kg/m^2 to <35 kg/m^2) at enrollment were evaluated at Week 16 to see if the same number who were obese at enrollment were still obese at Week 16 or if they had changed to an BMI of overweight (BMI of 25 kg/m^2 to <30 kg/m^2) or a BMI of normal (BMI of <25 kg/m^2) or a greater obesity (BMI >35 kg/m^2). Participants who were overweight (BMI of 25 kg/m^2 to <30 kg/m^2) at enrollment were evaluated at Week 16 to see if the same number who were overweight at enrollment were still overweight at Week 16 or if they had changed to normal (or obese).
Time Frame: Enrollment up to Week 16
Population: Evaluable: randomized participants with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with the protocol (per sponsor). Those excluded from Evaluable were identified prior to unblinding. Number analyzed were those participants with non-missing BMI data at enrollment and Week 16.
Measure: Number; unit: participants
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
participants
  Obese BMI at Enrollment | 14 | 30 | 27
  Continued Obese BMI at Week 16 | 9 | 11 | 11
  Decreased BMI to Overweight at Week 16 | 5 | 19 | 16
  Decreased BMI to Normal at Week 16 | 0 | 0 | 0
  Overweight BMI at Enrollment | 5 | 8 | 9
  Continued Overweight BMI at Week 16 | 4 | 8 | 5
  Decreased BMI to Normal at Week 16 | 1 | 0 | 4

13. Secondary Outcome: Number of Participants With BMI Change From Enrollment to Week 20 - Evaluable Population
Description: BMI was measured as kilogram per meter of height squared (kg/m^2). Enrollment was Visit 2 (Week -4). Participants who were obese (BMI of 30 kg/m^2 to <35 kg/m^2) at enrollment were evaluated at Week 20 to see if the same number who were obese at enrollment were still obese at Week 20 or if they had changed to an BMI of overweight (BMI of 25 kg/m^2 to <30 kg/m^2) or a BMI of normal (BMI of <25 kg/m^2) or a greater obesity (BMI >35 kg/m^2). Participants who were overweight (BMI of 25 kg/m^2 to <30 kg/m^2) at enrollment were evaluated at Week 20 to see if the same number who were overweight at enrollment were still overweight at Week 20 or if they had changed to normal (or obese).
Time Frame: Enrollment up to Week 20
Population: Evaluable: randomized participants with at least 1 dose of any treatment; completed Week 20 procedures and adequately complied with the protocol (per sponsor). Those excluded from Evaluable were identified prior to unblinding. Number analyzed were those participants with non-missing BMI data at enrollment and Week 20.
Measure: Number; unit: participants
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate+ Metreleptin
Number analyzed (Participants) | 19 | 37 | 36
participants
  Obese BMI at Enrollment | 14 | 29 | 27
  Continued Obese BMI at Week 20 | 7 | 10 | 10
  Greater Obesity at Week 20 | 1 | 0 | 0
  Decreased BMI to Overweight at Week 20 | 6 | 19 | 17
  Decreased BMI to Normal at Week 20 | 0 | 0 | 0
  Overweight BMI at Enrollment | 5 | 8 | 9
  Continued Overweight BMI at Week 20 | 4 | 8 | 5
  Decreased BMI to Normal at Week 20 | 1 | 0 | 4

14. Secondary Outcome: Mean Absolute Change From Enrollment to Week 16 in Fasting Glucose and Lipids - Evaluable Population
Description: Enrollment was Visit 2 (Week -4). Baseline refers to Visit 4 (Day 1 of randomization period). Fasting Lipids included: total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol, and Triglycerides. Fasting Glucose and Lipids were measured in milligrams per deciliter (mg/dL).
Time Frame: Enrollment to Week 16
Population: Evaluable: randomized participants with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with the protocol (per sponsor). Those excluded from Evaluable were identified prior to unblinding. n=number with non-missing data for lipids and glucose in each treatment group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
mg/dL
  Glucose (n=19, 35, 35) | -2.21 (8.574) | -1.86 (10.347) | -3.00 (7.412)
  Total Cholesterol (n=19, 38, 36) | 2.68 (25.164) | -10.76 (20.285) | -20.64 (25.798)
  HDL cholesterol (n=19, 38, 36) | 1.74 (6.358) | 1.63 (7.321) | -0.64 (7.761)
  LDL cholesterol (n=19, 38, 36) | 1.11 (22.266) | -5.50 (18.064) | -13.25 (17.986)
  Triglycerides (n=19, 37, 35) | 30.37 (77.920) | 1.57 (75.063) | -9.54 (53.844)

15. Secondary Outcome: Mean Absolute Change From Enrollment to Baseline, Weeks 4 and 16 in Fasting Total Leptin Concentration - Evaluable Population
Description: Enrollment was Visit 2 (Week -4). Baseline refers to Visit 4 (Day 1 of randomization period). Leptin was measured in nanograms per milliliter (ng/mL). Plasma total leptin (including endogenous leptin and exogenous metreleptin) concentrations were measured using a validated sandwich-type immunoenzymetric assay utilizing polyclonal capture antibody, monoclonal detection antibody, and colorimetric readout by Amylin Pharmaceuticals, Inc. This assay is not specific for metreleptin and detects both endogenous leptin and exogenous recombinant-methionyl human leptin [metreleptin]).
Time Frame: Enrollment to Week 16
Population: Evaluable: randomized participants with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with the protocol (per sponsor). Those excluded from Evaluable were identified prior to unblinding. n=number with non-missing data at visit in each treatment group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
ng/mL
  Baseline (Day 1) (n=18, 38, 35) | -6.16 (6.919) | -7.98 (6.932) | -7.23 (8.157)
  Week 4 (n=19, 38, 36) | 53.54 (98.124) | -6.56 (7.766) | 18.94 (38.475)
  Week 16 (n=19, 38, 36) | 375.28 (340.885) | -3.58 (13.296) | 262.61 (268.501)

16. Secondary Outcome: Mean Absolute Change From Enrollment to Baseline and Week 16 in Fasting Total Amylin -Evaluable Population
Description: Enrollment was Visit 2 (Week -4). Baseline refers to Visit 4 (Day 1 of randomization period). Fasting total plasma amylin (peptide produced by beta cells in the pancreas) concentration was measured in picomolar (pM) and samples were obtained at screening, enrollment, baseline, Week 4 and Week 16.
Time Frame: Enrollment to Week 16
Population: Evaluable: randomized participants with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with the protocol (per sponsor). Those excluded from Evaluable were identified prior to unblinding. n=number analyzed with non-missing data at visit.
Measure: Mean (Standard Deviation); unit: pM
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 18 | 37 | 36
pM
  Baseline (Day 1) (n=18, 37, 36) | -0.89 (4.258) | -2.18 (5.641) | -3.28 (4.378)
  Week 16 (n=18, 34, 36) | -3.31 (4.731) | -1.60 (5.720) | -2.17 (12.416)

17. Secondary Outcome: Mean Absolute Change From Enrollment to Baseline and Week 16 in Fasting Total Insulin - Evaluable Population
Description: Enrollment was Visit 2 (Week -4). Baseline refers to Visit 4 (Day 1 of randomization period). Total insulin was measured in micro international units per milliliter (µIU/mL)
Time Frame: Enrollment to Week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide + Metreleptin
Number analyzed (Participants) | 17 | 35 | 34
µIU/mL
  Baseline (Day 1) (n=17, 35, 34) | 0.00 (4.108) | -1.14 (4.095) | -0.68 (4.183)
  Week 16 (n=18, 34, 35) | -0.61 (4.877) | -0.65 (4.792) | -2.80 (3.385)

18. Secondary Outcome: LS Mean Absolute Change From Enrollment to Week 16 in Patient Reported Outcome (PRO) Instruments Measuring Quality of Life and Mood - Evaluable Population
Description: Enrollment was Visit 2 (Week -4). PRO: Total Score in Impact of Weight on Quality of Life Questionnaire-lite Version (IWQOL-Lite), 31-item instrument used to assess the effect of weight on physical function, self-esteem, sexual life, public distress, and work. Individual items range from 1 to 5 with 5=always true and 1= never true. Total score measured on scale from 0 (worst) to 100 (best). Higher scores indicate improvement; Profile of Mood States (POMS), 65 mood adjectives that assess participants' mood over the past seven days. The POMS-B is an authorized, 30-item brief version of the POMS consisting of five items for each: Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. Scores range from 0= Not at All to 4=Extremely. Factor scores added for total score. Lower score indicates improvement. 0=best outcome; 120=worst outcome.
Time Frame: Enrollment to Week 16
Population: Evaluable: randomized participants with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with the protocol (per sponsor). Those excluded from Evaluable were identified prior to unblinding. n=number with non-missing data at visit in each treatment group. (POMS)n=19, 38, 36; (IWQOL-Lite)n=19, 38, 36
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
units on a scale
  POMS Total Mood Disturbance Score(n=19, 38, 36) | -2.8 (6.17) | -4.5 (4.45) | -6.0 (4.50)
  IWQOL-Lite Total Score(n=19, 38, 36) | 12.14 (2.553) | 11.92 (1.843) | 12.49 (1.863)

19. Secondary Outcome: LS Mean Absolute Change From Enrollment to Week 16 in Patient Reported Outcomes (PRO) for Eating Behavior - Evaluable Population
Description: Enrollment was Visit 2 (Week -4). PRO for eating behavior: Binge Eating Scale (BES) Total Score (16-item questionnaire assessed the behavioral and cognitive correlates of binge eating, including participants' perceived self-control over eating behavior using a range of 1 to 4 with 1=positive perceptions and 4= negative perceptions. Minimum and maximum scores were 0 and 55, respectively); Susceptibility to Eating Questionnaire (SEQ) Total Score (measure of appetite, satiety, and perceived control over portion size using 10 VAS items with each response measured on a 100 mm visual analogue scale [ranges vary from Never to Very Often; Not at All Difficult to Extremely Difficult; Not at all Strong to Very Strong]. Responses to these items rated over the past 7 days;
Time Frame: Enrollment to Week 16
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
units on a scale
  BES Total Score (n=17, 36, 34) | -5.5 (1.27) | -3.8 (0.87) | -6.4 (0.89)
  SEQ Food Craving Frequency(n=19, 38, 36) | -21.8 (5.32) | -19.5 (3.84) | -24.6 (3.86)
  SEQ Strength of Food Cravings(n=19, 38, 36) | -16.8 (5.39) | -11.5 (3.88) | -19.8 (3.91)
  SEQ Difficult to Control Eating(n=19, 38, 36) | -23.0 (5.77) | -20.9 (4.17) | -29.3 (4.19)
  SEQ Difficult to Resist Food Cravings(n=19, 38, 36 | -22.7 (5.47) | -18.6 (3.95) | -30.2 (3.97)
  SEQ Response to Food Cravings(n=19, 38, 36) | -22.0 (5.30) | -22.6 (3.83) | -33.4 (3.85)
  SEQ Control Portion Sizes(n=19, 38, 36) | -24.8 (5.26) | -27.5 (3.78) | -33.1 (3.78)
  SEQ How Hungry(n=19, 38, 36) | -21.1 (5.20) | -18.5 (3.77) | -28.5 (3.77)
  SEQ How Full After Meal(n=19, 38, 36) | -3.0 (5.20) | 2.8 (3.76) | -4.6 (3.77)
  SEQ Thoughts of Food(n=19, 38, 36) | -20.4 (5.62) | -11.6 (4.07) | -21.5 (4.07)
  SEQ How Pleasant Meals(n=19, 38, 36) | -3.2 (4.73) | -0.8 (3.42) | -6.5 (3.44)

20. Secondary Outcome: LS Mean Absolute Change From Enrollment to Week 16 in Hospital Anxiety and Depression Scale (HADS) - Evaluable Population
Description: The HADS is a questionnaire that uses 14 items to assess both anxiety and depression over the past week. The odd numbered items constitute the anxiety subscale, and the even numbered items constitute the depression subscale. The individual response scores for each subscale component are added together to obtain the individual subscale scores. The minimum and maximum score for each subscale is 0 and 21, respectively. The lower the score the more improvement a participant shows.
Time Frame: Enrollment to Week 16
Population: Evaluable: randomized participants with at least 1 dose of any treatment; completed Week 16 procedures and adequately complied with the protocol (per sponsor). Those excluded from Evaluable were identified prior to unblinding. Number with non-missing data in each treatment group were analyzed (n).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 38 | 36
units on a scale
  Anxiety Total (n=19, 38, 36) | -0.7 (0.71) | -0.1 (0.51) | -0.3 (0.51)
  Depression Total (n=19, 38, 36) | -0.7 (0.56) | -0.5 (0.40) | -0.5 (0.40)

21. Secondary Outcome: Mean Absolute Change From Enrollment to Week -2, Week 16 and Week 20 in Systolic and Diastolic Blood Pressure - Enrolled Population
Description: Enrollment was Visit 2 (Week -4). Blood pressure (BP) was measured after 5 minutes of quiet rest with the participant in a sitting position and was measured in millimeters of mercury (mm Hg). Blood pressure was taken at each visit (screening, Week -4, Week -2, Day 1, Weeks 4, 8, 12, 16, 20 (or early termination). After the Lead-In Period, participants were either randomized to one of the 3 arms of the study or they were dropped from the study so the time frame for evaluation of all participants in the study was either: enrollment up to Week 20 for Randomized participants or enrollment up to, but not including Day 1 for Non-Randomized participants who participated only in the Lead-In Period.
Time Frame: Enrollment up to Week 20(Randomized Group) or Enrollment up to, not including Day 1(Non-Randomized Group)
Population: ITT:those randomized, received at least 1 injection of any component of the randomized medication. Enrolled not randomized: those who received at least 1 dose of pramlintide in 4-week lead-in period. n=number with non-missing data at visit in each treatment group.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin | Non-Randomized From 4 Week Lead-In
Number analyzed (Participants) | 27 | 56 | 56 | 38
mm Hg
  Systolic BP Change up to Week -2(n=27,56,56,23) | -1.2 (8.06) | -3.5 (8.74) | -2.8 (9.08) | 0.9 (9.94)
  Diastolic BP Change up to Week -2(n=27,56,56,23) | -3.7 (6.10) | -1.8 (6.51) | -1.9 (7.06) | -0.6 (6.08)
  Systolic BP Change to Week 16(n=19,39,38) | -6.3 (7.98) | -4.5 (9.41) | -1.6 (10.06) | NA (NA) — Non-randomized participants (total of 38) are those who left the study before being randomized to a treatment group. These 38 participants received pramlintide in the Lead-In Period.
  Diastolic BP Change to Week 16(n=19,39,38) | -3.7 (6.88) | -2.6 (7.16) | 0.3 (8.57) | NA (NA) — Non-randomized participants (total of 38) are those who left the study before being randomized to a treatment group. These 38 participants received pramlintide in the Lead-In Period.
  Systolic BP Change to Week 20(n=19,37,38) | -1.2 (11.28) | -3.9 (9.64) | -1.9 (8.76) | NA (NA) — Non-randomized participants (total of 38) are those who left the study before being randomized to a treatment group. These 38 participants received pramlintide in the Lead-In Period.
  Diastolic BP Change to Week 20(n=19,37,38) | -1.5 (8.12) | -1.0 (8.15) | 1.8 (7.59) | NA (NA) — Non-randomized participants (total of 38) are those who left the study before being randomized to a treatment group. These 38 participants received pramlintide in the Lead-In Period.

22. Secondary Outcome: Absolute Change From Enrollment to Week -2, Week 16 and Week 20 in Heart Rate - Enrolled Population
Description: Enrollment was Visit 2 (Week -4). Heart rate was measured after the participant rested for 5 minutes and was sitting. Heart Rate was measured in beats per minute (bpm). Vital signs were taken at each visit (screening, Week -4, Week -2, Day 1, Weeks 4, 8, 12, 16, 20 (or early termination). After the Lead-In Period, participants were either randomized to one of the 3 arms of the study or they were dropped from the study so the time frame for evaluation of all participants in the study was either: enrollment up to Week 20 for Randomized participants or enrollment up to, but not including Day 1 for Non-Randomized participants who participated only in the Lead-In Period.
Time Frame: Enrollment up to Week 20(Randomized Group) or Enrollment up to, not including Day 1(Non-Randomized Group)
Population: ITT: those randomized, received at least 1 injection of any component of the randomized medication. Enrolled not randomized: those who received at least 1 dose of pramlintide in 4-week lead-in period. n=number with non-missing data at visit in each treatment group.
Measure: Mean (Standard Deviation); unit: beats/min
Groups:
- Non-Randomized From 4 Week Lead-In: During the 4-week lead-in period, all participants self administered subcutaneous (SC) injections of pramlintide acetate180 mcg twice per week (BID) for 2 weeks followed by pramlintide acetate 360 mcg BID for 2 weeks while following a diet aimed at creating a 40% caloric deficit relative to their estimated weight-maintenance energy needs. Participants who lost between 2% and 8% of their enrollment body weight during the lead-in period were randomized at Visit 4 (baseline/Day 1) to 1 of 3 treatment groups (metreleptin, pramlintide, or pramlintide+metreleptin). 38 participants were not randomized into one of the 3 treatment groups and withdrew from the study.
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin | Non-Randomized From 4 Week Lead-In
Number analyzed (Participants) | 27 | 56 | 56 | 38
beats/min
  Week -2 (n=27,56,56,23) | -1.3 (10.76) | -0.8 (7.82) | -1.1 (8.83) | 1.3 (12.05)
  Week 16 (n=19, 39, 38) | -0.2 (11.09) | -2.1 (7.58) | -4.2 (9.47) | NA (NA) — Non-randomized participants (total of 38) are those who left the study before being randomized to a treatment group. These 38 participants received pramlintide in the Lead-In Period.
  Week 20 (n=19, 37, 38) | -0.2 (8.90) | -1.6 (6.50) | -3.8 (10.21) | NA (NA) — Non-randomized participants (total of 38) are those who left the study before being randomized to a treatment group. These 38 participants received pramlintide in the Lead-In Period.

23. Secondary Outcome: Number of Chemistry Values of Potential Clinical Importance - Enrolled Population
Description: Number of values (not participants). Greater than (>), Less than (<), high (H), low (L). Criteria for laboratory values of potential clinical importance for obese and overweight (BMI>=25 kg/m^2) participants: Total bilirubin H > 2 mg/dL; glucose fasting or non-fasting H >200 mg/dL, L <60 mg/dL; Albumin L <2.5 g/dL; Creatine Phosphokinase (CPK) H >3*Upper limit of Normal (ULN); Sodium L<130 milliequivalents per liter (mEq/L), H >150 mEq/L; potassium L<3.0 mEq/L, H>5.5 mEq/L;bicarbonate L<18 mEq/L, H>35 mEq/L;calcium L <8 mg/dL, H>11 mg/dL; triglycerides H>500 mg/dL; Cholesterol L < 100 mg/dL, H > 350 mg/dL; Alkaline phosphatase H >3*ULN; Gamma-glutamyltransferase (GGT) H>3*ULN; creatinine males >1.6 mg/dL, females >1.4 mg/dL; alanine aminotransferase (ALT) H >3*ULN; aspartate aminotransferase (AST) H >3*ULN; urea nitrogen H >45 mg/dL; uric acid males >10.0 mg/dL, females > 8.0 mg/dL; Phosphorus L <1.0 mg/dL H >6.0 mg/dL. Time frame differs depending on randomization status.
Time Frame: Enrollment up to Week 20(Randomized Group) or Enrollment up to, not including Day 1(Non-Randomized Group)
Population: The Enrolled Population includes all enrolled participants who received at least 1 dose of pramlintide during the 4-week lead-in period or who had nonmissing data at Week -4. n=number with non-missing data in each treatment group who were in the analysis.
Measure: Number; unit: laboratory values
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin | Non-Randomized From 4 Week Lead-In
Number analyzed (Participants) | 27 | 56 | 56 | 37
laboratory values
  ALT (n=27, 56, 56, 37) | 0 | 1 | 0 | 0
  AST (n=27, 56, 56, 37) | 0 | 1 | 0 | 0
  Bicarbonate (n=27, 55, 56, 37) | 3 | 7 | 4 | 0
  CPK (n=27, 56, 56, 37) | 0 | 1 | 6 | 0
  GGT (n=27, 56, 56, 37) | 1 | 2 | 0 | 0
  Phosphorus (n=27, 56, 56, 37) | 0 | 0 | 0 | 1
  Potassium (n=27, 56, 56, 37) | 0 | 1 | 0 | 2
  Sodium (n=27, 56, 56, 37) | 0 | 1 | 0 | 0
  Total bilirubin (n=27, 56, 56, 37) | 0 | 1 | 0 | 0
  Triglycerides (n=27, 56, 56, 37) | 1 | 0 | 0 | 0
  Uric Acid (n=27, 56, 56, 37) | 1 | 0 | 0 | 0

24. Secondary Outcome: Number of Hematology and Urinalysis Values of Potential Clinical Importance - Enrolled Population
Description: Number of laboratory values of potential clinical importance (not participants) observed. Criteria for laboratory values of potential clinical importance for obese and overweight (BMI >= 25 kg/m^2) participants: Platelets high (H) >500,000/µL; low (L) <75,000/µL. Hematocrit males <36%, females <30%. Hemoglobin males <12 g/dL, females <10 g/dL. White blood cell count (WBC) H >18,000/µL; L <1,500/µL. Urine protein H >= 3+ or >= 500 mg/dL. Urine glucose H >= 3+ or >= 500 mg/dL. Urine ketones >= 3+ or Large. Time frame of evaluation differs depending on randomization status.
Time Frame: Enrollment up to Week 20(Randomized Group) or Enrollment up to, not including Day 1(Non-Randomized Group)
Population: The Enrolled Population includes all enrolled participants who received at least 1 dose of pramlintide during the 4-week lead-in period or who had nonmissing vital signs data at Week -4. n=number with non-missing data in each treatment group
Measure: Number; unit: participants
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin | Non-Randomized From 4 Week Lead-In
Number analyzed (Participants) | 27 | 56 | 56 | 38
participants
  Hematocrit (n=27, 55, 54, 35) | 0 | 3 | 1 | 0
  Hemoglobin (n=27, 56, 54, 36) | 0 | 2 | 1 | 0
  Urine Protein Positive (n=27, 56, 56, 37) | 0 | 1 | 4 | 0

25. Secondary Outcome: Number of Participants With Clinically Significant Abnormal ECG at Weeks 16, 20, or Early Termination - Randomized Population
Description: A 12-Lead electrocardiogram (ECG) was obtained at Week -4, Day 1, Week 16, Week 20 or early termination and the overall interpretation of the ECG was made by the investigator as normal, abnormal (not clinically significant) and abnormal (clinically significant). The ECG consisted of the PR interval = time from beginning of the P wave to the beginning of the QRS complex; (Note: QRS complex is a name for the combination of 3 of the graphical deflections seen in an ECG); QRS (time from the beginning to the end of the QRS complex) interval; QT interval (measure between Q wave and T wave in the heart's electrical cycle); and QT interval corrected for heart rate using Fridericia's formula (QTcF) were measured in milliseconds (msec). .
Time Frame: Weeks 16, 20, early termination
Population: All participants who were enrolled and randomized and had ECGs performed at Weeks 16, 20, or early termination. n=number of participants with ECGs at visit by treatment group.
Measure: Number; unit: participants
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 19 | 39 | 38
participants
  Week 16 (n=19, 39, 38) | 0 | 0 | 0
  Week 20 (n=19, 37, 37) | 0 | 0 | 0
  Early Termination (n=4, 6, 11)) | 0 | 0 | 0

26. Secondary Outcome: Number of Participants With Treatment-emergent Anti-Leptin Antibodies by Week 4, Week 8, Week 12, Week 16 - Intent to Treat Population
Description: Serum titer determinations for antibodies to leptin were made using a validated electrochemical luminescence (ECLA) bridging assay. Antibody titers were assessed according to the following dilutions: 0, 5, 25, 125, 625, 3125, 15625, and 78125. Participants were considered to have a positive titer to treatment-emergent antibodies to leptin at a given visit if they had a titer >=5 following a negative or missing titer at baseline or if they had a titer that had increased by at least 2 dilutions from a detectable level at baseline. All participants were evaluated (including those who did not receive metreleptin as their randomized study drug). Baseline was Day 1 (randomization).
Time Frame: Baseline up to Week 16
Population: The Intent-To-Treat (ITT) Population includes all randomized participants who received at least 1 injection of any component of the randomized study medication; n=number with non-missing data at visit in each treatment group.
Measure: Number; unit: participants
Arm/Group | Metreleptin | Pramlintide Acetate | Pramlintide Acetate + Metreleptin
Number analyzed (Participants) | 22 | 48 | 45
participants
  Week 4 (n=22, 48, 45) | 19 | 3 | 39
  Week 8 (n=19, 46, 37) | 19 | 0 | 37
  Week 12 (n=19, 40, 38) | 19 | 0 | 38
  Week 16 (n=19, 38, 38) | 19 | 1 | 38

ADVERSE EVENTS:
Time Frame: 4 Week Lead-in Period and 20 weeks Randomized Treatment Period (24 weeks total)
Description: systematic assessment for administration site adverse events and non-systematic assessment for all other adverse events.
Groups:
- Placebo + Metreleptin: Participants self administered subcutaneous (SC) injections of Placebo matched to pramlintide (Placebo-P) BID plus Metreleptin 5 mg BID. Dosing for up to 20 weeks. Participants were asked to maintain a 20% caloric deficit during the treatment period.
- Pramlintide + Placebo: Participants self administered subcutaneous (SC) injections of Pramlintide 360 mcg BID plus Placebo matched to Metreleptin (Placebo-M) BID. Dosing for up to 20 weeks. Participants were asked to maintain a 20% caloric deficit during the treatment period.
- Participants Not Randomized to Group After Lead-In Period: During the 4-week lead-in period, all participants self administered a subcutaneous injection of pramlintide 180 mcg twice per week (BID) for 2 weeks followed by pramlintide 360 mcg BID for 2 weeks while following a diet aimed at creating a 40% caloric deficit relative to their estimated weight-maintenance energy needs. Participants who lost between 2% and 8% of their enrollment body weight during the lead-in period were randomized at Visit 4 (baseline/Day 1) to 1 of 3 treatment groups (metreleptin, pramlintide, or pramlintide+metreleptin). 38 participants were not Randomized into one of the 3 treatment groups and withdrew from the study.
Arm/Group | Placebo + Metreleptin | Pramlintide + Placebo | Pramlintide + Metreleptin | Participants Not Randomized to Group After Lead-In Period
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/56 | 2/56 | 0/38
Other Adverse Events (participants affected / at risk) | 24/27 | 42/56 | 45/56 | 17/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Metreleptin (N=27) | Pramlintide + Placebo (N=56) | Pramlintide + Metreleptin (N=56) | Participants Not Randomized to Group After Lead-In Period (N=38)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Metreleptin (N=27) | Pramlintide + Placebo (N=56) | Pramlintide + Metreleptin (N=56) | Participants Not Randomized to Group After Lead-In Period (N=38)
Injection Site Bruising (General disorders) | 3 (3) | 9 (11) | 11 (13) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 8 (10) | 7 (8) | 10 (10)
Injection Site Erythema (General disorders) | 5 (5) | 6 (8) | 8 (8) | 0 (0)
Injection Site Pruritus (General disorders) | 7 (7) | 3 (3) | 8 (8) | 0 (0)
Injection Site Urticaria (General disorders) | 5 (5) | 0 (0) | 9 (10) | 0 (0)
Injection Site Nodule (General disorders) | 4 (4) | 3 (3) | 3 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 7 (7) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 4 (5) | 3 (4) | 1 (1)
Injection Site Haemorrhage (General disorders) | 1 (2) | 6 (7) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (3) | 2 (3)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Injection Site Induration (General disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Injection Site Rash (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.